CLINICAL TRIAL: NCT05315401
Title: The Efficacy of Probiotic Compared With Placebo and Acceptance and Commitment Therapy for the Treatment of Major Depressive Disorder Among Adult Females
Brief Title: The Efficacy of Probiotic Compared With Placebo Commitment Therapy for Treatment of Major Depressive Disorder
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Fail to recruit
Sponsor: Min-Tze LIONG (Other)
Collaborators: National University of Malaysia (Other)
Responsible Party: Sponsor-Investigator, Min-Tze LIONG, Professor.Dr, Universiti Sains Malaysia
Organization: Universiti Sains Malaysia (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: JEP-2021-606
Record Dates: First submitted 2022-03-30; First posted 2022-04-07 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Major Depressive Disorder
Keywords: Probiotics
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Probiotics; Acceptance and Commitment Therapy

STUDY DESIGN:
Intervention Model Description: A double-blind three-armed randomized controlled trial design has been chosen. Randomization for the parallel prevention phase will be carried out after checking the inclusion and exclusion criteria
Who Masked: Participant, Care Provider, Investigator
Masking Description: . The randomization will be performed by the study statistician, who had no contact with the patients and not involve in the research project. The allocation sequence will not be available to any member of the research team until databases had been completed and locked. Since this is a double-blinded study, both the research team and subject will not know in which group the subject is assigned to.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Probiotic 9 log CFU/day (Experimental): The intervention consists of daily administration of one sachet/day of probiotic for 12 weeks, where each sachet contains 9 log CFU of probiotic.
  Interventions: Dietary Supplement: Probiotic
- Placebo (Placebo Comparator): placebo contains primarily carrier and without probiotic. The placebo are identical in taste and appearance and appear as a light-yellow powder.
  Interventions: Dietary Supplement: Placebo
- Acceptance and commitment therapy (ACT) (Experimental): Patients will be provided with ACT for 12 weeks with treatment as usual. The ACT intervention will be conducted in a group of 10 for each session. The ACT modules covered over 12 sessions, 1 hour in each session. The sessions will be held every week
  Interventions: Behavioral: Acceptance and commitment therapy (ACT)

INTERVENTIONS:
Dietary Supplement: Probiotic — This project aims to evaluate the efficacy of oral administration of probiotic at 9 log CFU/day as adjunctive treatment in reducing the severity depression in female patients with major depressive disorder with treatment-as-usual compared to placebo and ACT via use of questionnaires.
  Arms: Probiotic 9 log CFU/day
Dietary Supplement: Placebo — This project aims to evaluate the efficacy of oral administration of probiotic at 9 log CFU/day as adjunctive treatment in reducing the severity depression in female patients with major depressive disorder with treatment-as-usual compared to placebo and ACT via use of questionnaires.
  Arms: Placebo
Behavioral: Acceptance and commitment therapy (ACT) — Patients will be provided with ACT for 12 weeks with treatment as usual. The ACT intervention will be conducted in a group of 10 for each session. The ACT modules covered over 12 sessions, 1 hour in each session. The sessions will be held every week.
  Arms: Acceptance and commitment therapy (ACT)

SUMMARY:
The purpose of this study is to evaluate the efficacy of oral administration of probiotic at 9 log CFU/day as adjunctive treatment in reducing the severity of depression in female patients with major depressive disorder with treatment-as-usual compared to placebo and ACT via the use of questionnaires.

DETAILED DESCRIPTION:
1. To assess the differences in quality of life among patients on probiotic, placebo and ACT via the use of questionnaire, at 4 timelines (baseline, 6 weeks after starting intervention, 12 weeks after starting intervention, and 24 weeks after starting intervention which is 12 weeks post-termination of intervention).
2. To assess the differences in blood biological markers such as BDNF, TNF-α, IL-6, IL-1β, CRP, and VEGF among patients on probiotic, placebo and ACT via blood biochemical analyses, at 4 timelines (baseline, 6 weeks after starting intervention, 12 weeks after starting intervention, and 24 weeks after starting intervention which is 12 weeks post-termination of intervention).
3. To assess the differences in gut microbiota profiles of patients on probiotic, placebo and ACT via the use of fecal samples, at 3 timelines (baseline, 12 weeks after starting intervention, and 24 weeks after starting intervention which is 12 weeks post-termination of intervention).

ELIGIBILITY:
Inclusion Criteria:

* Female patient diagnosed with major depressive disorder (confirmed by DSM-5 for depression). There is a strong gender predisposition in depression and anxiety disorders, in which females are more prone to have depressive disorders and anxiety disorders than males. Hence, we will only recruit female patients in this study to control for confounding bias.
* Those with score of more than 8 based on Hamilton Depression Rating Scale (HAMD), indicative of mild to moderate severity of depressive symptoms.
* Age 18 to 35 years old

Exclusion Criteria:

* Pregnant women
* Those who have current and lifetime history of engaging in any psychotherapy
* Those who consumed alcohol and illicit drugs (Heavy or mild)
* Those who has current and lifetime history of other psychiatric illnesses, such as other depressive disorders (persistent depressive disorder, premenstrual dysphoric disorder), anxiety disorders (panic disorder, agoraphobia, generalized anxiety disorder, specific anxiety disorder, and social anxiety disorder), psychotic disorders (schizophrenia, schizophreniform disorder, schizoaffective disorders, brief psychotic disorder, and delusional disorder), bipolar mood disorder, obsessive compulsive disorder, posttraumatic stress disorder, and attention deficit hyperactive disorder, and autism spectrum disorder
* Those who are on medications that can induce psychiatric symptoms, such as cardiovascular agents (clonidine, guanethidine, methyldopa, reserpine, beta blockers), dermatologic agents (isotretinoin), anticonvulsants (levetiracetam), antimigraine medications (triptans), hormonal agents (corticosteroids, oral contraceptives, gonadotropin-releasing hormone agonists, tamoxifen), varenicline, immunological agents (interferons), and levodopa
* Severe gastritis with regular intake omeprazole medication (proton pump inhibitors)
* Women on regular steroid treatment
* Those on long term medication for any illnesses (≥ 6 months)
* Those who are currently on antibiotics or with history of taking antibiotic for the past 2 weeks.
* Those with abnormal full blood count, renal profile, liver function test, fasting blood glucose, fasting lipid profile and ESR (blood collection for all these blood investigations will be carried out in the pre-intervention assessment).
* Patient who has suicidal tendency

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
differences in severity of depression in patients with major depressive disorder upon consumption of probiotic at 9 log CFU/day compared to placebo and ACT. | 24 weeks
  To evaluate differences in severity of depression via the use of the Montgomery and Åsberg (MADRS) Depression Rating Scale questionnaire containing 10-items on a 7-point scale with higher scores indicating more severe depression

SECONDARY OUTCOMES:
differences in quality of life in patients with major depressive disorder upon consumption of probiotic at 9 log CFU/day compared to placebo and ACT. | 24 weeks
  To evaluate differences in quality of life via the use of the RAND-36 questionnaire containing 36-items on a varying point scale including some items with reverse scoring, with higher scores indicating better health status.
differences in blood depression biomarkers in patients with major depressive disorder upon consumption of probiotic at 9 log CFU/day compared to placebo and ACT. | 24 weeks
  To evaluate differences in depression blood biological markers such as BDNF, TNF-α, IL-6, IL-1β, CRP, and VEGF via measuring concentrations using commercially available ELISA kit.
differences in gut microbiota profiles of patients with major depressive disorder upon consumption of probiotic at 9 log CFU/day compared to placebo and ACT. | 24 weeks
  To evaluate differences in gut microbiota profiles via microbiota profiling using DNA of fecal samples amplified for bacterial 16S rRNA and analyzed for high-throughput community sequencing.

CONTACTS AND LOCATIONS:
Overall Officials: Min Tze Liong, Prof.Dr, Study Director — School of Industrial Technology, University of Science Malaysia; Luke Woon Sy-Cherng, Dr, Principal Investigator — Department of Psychiatry Hospital Canselor Tuanku Muhriz UKM medical Centre
Locations (1):
- Hospital Canselor Tuanku Muhriz UKM Medical Centre, Cheras, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No